CLINICAL TRIAL: NCT02895256
Title: Long-term Prognosis of Cluster Headache: a Retrospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Chin-Sang Chung, MD, PhD, Professor of neurology, Samsung Medical Center
Other Study IDs: 2016-04-155
Record Dates: First submitted 2016-09-04; First posted 2016-09-09 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Cluster Headache; Disease Course
MeSH Terms: conditions — Cluster Headache; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Any treatment for cluster headache

SUMMARY:
Cluster headache is a syndrome characterized by disabling headache and accompanying autonomic symptoms. Despite cluster headache is called "suicide headache", its natural history has not been well investigated. The investigators aimed to investigate its disease course, overall prognosis, and treatment pattern in retrospective cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed as cluster headache
* More than 5 years after the first visit

Exclusion Criteria:

* Subjects who refused the telephone visit

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cluster headache
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2016-04; Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
overall prognosis | at least 5 years after the first visit
  active disease: at least one bout within the past 5 years Remission: no headache for 5 years and twice of the usual remission period
Changes in the length of active/inactive periods | at least 5 years after the first visit
Changes in seasonal and diurnal predilections | at least 5 years after the first visit
Changes in autonomic symptoms | at least 5 years after the first visit
Changes in treatment responses | at least 5 years after the first visit

SECONDARY OUTCOMES:
Any depression | at least 5 years after the first visit
Any suicidal thoughts (active/passive), plans, and attempts | at least 5 years after the first vis
  ictal vs interictal

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea